CLINICAL TRIAL: NCT04372615
Title: A Phase-2b, Double-Blind, Randomized Controlled Trial to Evaluate the Activity and Safety of Inebilizumab in Anti-Nmda Receptor Encephalitis and Assess Markers of Disease
Brief Title: The ExTINGUISH Trial of Inebilizumab in NMDAR Encephalitis
Acronym: ExTINGUISH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Stacey Clardy MD PhD, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 143461
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Autoimmune Encephalitis; Encephalitis
Keywords: Inebilizumab; NMDAR encephalitis; Autoimmune Encephalitis; Rare Disease
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Encephalitis; Rare Diseases | interventions — inebilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inebilizumab (Active Comparator): Approximately 58 patients will receive Inebilizumab in addition to first line immunotherapy.
  (Approximately 116 participants will be randomized in a 1:1 ratio to 2 treatment groups; approximately 58 participants to each treatment group).
  All participants will also receive a 3 day course of IVIg.
  Interventions: Drug: Inebilizumab
- Placebo (Placebo Comparator): Approximately 58 patients will receive placebo in addition to first line immunotherapy.
  (Approximately 116 participants will be randomized in a 1:1 ratio to 2 treatment groups; approximately 58 participants to each treatment group).
  All participants will also receive a 3 day course of IVIg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inebilizumab — RCP: Blinded treatment on Day 1, Day 15,
  * Inebilizumab group: Inebilizumab 300 mg intravenous (IV)
  * Placebo group: IV matching placebo Prior to enrollment, all participants will receive standard of care, including high-dose corticosteroids (minimum of 3 days of treatment, 1 g methylprednisolone daily or equivalent) AND either IVIg (total dose range between 1.2 and 2 g/kg) OR plasmapheresis (defined as 5 or 6 exchanges).
  Rescue therapy will be given to participants in either treatment group based on the results of the Week 6 assessments. Rescue therapy is cyclophosphamide 750 mg/m2 IV followed by additional doses every 28-30 days until the mRS score is ≤ 3 (at site Principal Investigator's discretion under standard of care).
  Other Names: UPLIZNA
  Arms: Inebilizumab
Drug: Placebo — The placebo group will receive IV matching placebo on Day 1 and Day 15,
  Arms: Placebo

SUMMARY:
Determine the difference in the modified Rankin score at 16 weeks in participants with anti-N-methyl-D-aspartate receptor (NMDAR) encephalitis treated with "first-line" immunomodulatory therapies provided as standard-of-care, and either inebilizumab (investigational agent) or placebo.

DETAILED DESCRIPTION:
N-methyl-D-aspartate receptor (NMDAR) encephalitis is one of the most common causes of autoimmune encephalitis, with prevalence exceeding herpes encephalitis in industrialized nations. Typically, the disease affects patients age 10-50 causing prominent psychiatric symptoms, altered consciousness, seizures, movement disorders and life-threatening dysautonomia. Intensive care, including cardiorespiratory support is required in 75% of cases. The diagnosis is confirmed by detection of IgG autoantibodies against central nervous system NMDAR in the cerebrospinal fluid. Despite the severity of the illness, NMDAR encephalitis is a treatable neurological disease, with retrospective case series establishing the benefit of off-label intravenous steroids and immunoglobulins. These treatments are presumed to work through effects on IgG NMDAR autoantibody levels in the CSF, although prospective data informing predictors of treatment responses are limited. Even with prompt treatment, ~50% of patients remain disabled, requiring prolonged hospital admissions. Various off-label therapies have been proposed as "second-line" treatments in NMDAR encephalitis. The majority of second-line treatments target circulating B-cells with various degrees of blood brain penetrance and efficacy, and poor consensus on the timing, dose and route of delivery of candidate agents. High-quality evidence is needed to inform the treatment of NMDAR encephalitis. Inebilizumab is a promising therapeutic monoclonal antibody for the treatment of NMDAR encephalitis. This humanized monoclonal antibody against the B-cell surface antigen CD19 was recently shown to be safe and efficacious in the treatment of neuromyelitis optica spectrum disorder-another antibody-mediated disorder of the central nervous system. Compared to other off label B-cell depleting therapies, such as rituximab, inebilizumab not only depletes CD20+ B-cells, but also CD20- plasmablasts and plasma cells, resulting in robust and sustained suppression of B-cell expression. The ExTINGUISH Trial will randomize 116 participants with moderate-to-severe NMDAR encephalitis to receive either inebilizumab or placebo in addition to first-line therapies. Patient outcomes will be ascertained at standard intervals using the modified Rankin scale and accepted safety measures (primary outcomes at 16 weeks), together with comprehensive validated neuropsychological tests, bedside cognitive screening tools, quality of life/ functional indices, and outcome prediction measures. Clinical data will be combined with quantitative measures of NMDAR autoantibody titers and cytokines implicated in B-cell activation and antibody production within the intrathecal compartment to identify treatment responders, inform the biologic contributors to outcomes, and evaluate for biomarkers that may serve as early predictors of favorable outcomes in future clinical trials in NMDAR encephalitis. The ExTINGUISH Trial will prospectively study an optimized B-cell depletion therapy to promote better long-term outcomes in NMDAR encephalitis, to determine more meaningful cognitive endpoints, and to identify better biologic biomarkers to predict outcome.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of NMDAR encephalitis, defined by both a and b:

   1. A subacute onset of change in mental status consistent with autoimmune encephalitis,
   2. A positive cell-based assay for anti-NMDA receptor IgG antibody in the CSF confirmed in study-specified laboratories.
2. Participants, ≥ 12 years of age at the time of informed consent. Participants under 18 years of age must weigh ≥40 kilograms.
3. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA] in the United States of America [USA], European Union [EU] Data Privacy Directive in the EU) obtained from the participant/legal representative prior to performing any protocol-related procedures, including screening evaluations.
4. Non-sterilized participants who are sexually active with a partner capable of becoming pregnant must use a condom with spermicide from Day 1 through to the end of the study and must agree to continue using such precautions for at least 6 months after the final dose of IP. A recommendation will be made that the partners (capable of becoming pregnant) of study participants (capable of getting their partner pregnant) should use a highly effective method of contraception other than a physical method.

   Participants of childbearing potential who are sexually active with a non-sterilized partner capable of getting their partner pregnant must agree to use a highly effective method of contraception beginning at screening or upon discharge from hospitalization/inpatient rehabilitation (for participants who were incapacitated at the time of screening), and to continue precautions for 12 months after the final dose of IP.
   1. Participants of childbearing potential are defined as those who are not surgically sterile (e.g., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are not postmenopausal (per ICH M3 (R2) 11.2: defined as 12 months with no menses without an alternative medical cause).
   2. A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Periodic abstinence, the rhythm method, and the withdrawal method do not qualify as "highly effective" or acceptable methods of contraception for study purposes. Acceptable methods of contraception are listed in the table below:

      Physical Methods Hormonal Methods e

      • Intrauterine device (IUD)

      • Intrauterine hormone-releasing system, also known as drug-eluting IUD a

      • Bilateral tubal occlusion

      • Vasectomized partner b

      • Sexual abstinence c • Combined (estrogen and progestogen-containing hormonal contraception)
      * Oral (combined pill)
      * Injectable
      * Transdermal (patch)
      * Progestogen-only hormonal contraception associated with inhibition of ovulation d
      * Implantable
      * Intravaginal a This is also considered to be a hormonal method. b With appropriate post-vasectomy documentation of surgical success (absence of sperm in ejaculate).

      c Sexual abstinence is considered to be a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of the study and if it is the preferred and usual lifestyle of the participant.

      d Progestogen-only hormonal contraception, where inhibition of ovulation is not the primary mode of action (minipill) is not accepted as a highly effective method.

      e These methods are only considered highly effective and therefore acceptable when used in conjunction with a barrier method (i.e., diaphragm with spermicide, sponge with spermicide, cervical cap with spermicide, condoms, spermicide alone.)
5. Willing to forgo other immunomodulatory therapies (investigational or otherwise) for NMDAR encephalitis during the study.
6. Participant must have received at least 3 days of methylprednisolone 1000 mg IV or equivalent corticosteroid within 90 days prior to randomization (Day 1). In addition, participants must have received EITHER of the following treatments within 90 days before randomization.

   1. IVIg, at a dose range between 1.2 and 2 g/kg
   2. Plasma exchange or plasmapheresis, (defined as 5 to 6 exchanges).

   NOTE: These treatments may be provided during the screening period but must be completed prior to randomization. Participants who receive methylprednisolone and BOTH IVIg and plasma exchange are not excluded from participating in the trial, however, this treatment course with both IVIg and plasma exchange is not encouraged, and enrollment and randomization should not be delayed in order to complete additional first line treatments.
7. Modified Rankin Score of ≥3 at the screening visit, indicating at least moderate disability. The baseline mRS must be confirmed by Site Investigators at screening and confirmed / adjudicated before randomization.
8. Ability and willingness to attend study visits and complete the study. *All inclusion criteria must be met during the screening period, prior to randomization, except where noted.

Exclusion Criteria

Any of the following excludes an individual from participation in the study:

1. Any condition that, in the opinion of the Investigator, would interfere with the evaluation or administration of the IP, interpretation of participant safety or study results, or would make participation in the study an unacceptable risk. This specifically includes recent history (last 5 years) of herpes simplex virus encephalitis or known central nervous system demyelinating disease (e.g., multiple sclerosis).
2. Presence of an active or chronic infection that is serious in the opinion of the Investigator.
3. History of solid organ or cell-based transplantation.

<!-- -->

1. Concurrent/previous enrollment in another clinical study involving an investigational treatment within 4 weeks or 5 published half-lives of the investigational treatment, whichever is longer, prior to randomization.
2. Lactating or pregnant individuals, or individuals who intend to become pregnant anytime from study enrollment to 12 months following last dose of investigational agent.
3. Known history of allergy or reaction to any component of the investigational agent formulation or history of anaphylaxis following any biologic therapy.
4. Receipt of the following at any time prior to randomization:

   a. Alemtuzumab b. Total lymphoid irradiation c. Bone marrow transplant d. T-cell vaccination therapy
5. Receipt of any biologic B cell-depleting therapy (e.g., rituximab, ocrelizumab, obinutuzumab, ofatumumab, inebilizumab) in the 6 months prior to screening. Receipt of such a B cell-depleting agent in the period 6-12 months prior to screening is exclusionary unless B cell counts have returned to ≥ age-based LLN by central laboratory. For EU participants, B cell counts at screening will be determined by the laboratories of the participating sites. Receipt of non-depleting B cell-directed therapy (e.g., belimumab), abatacept, or other biologic immunomodulatory agent within 6 months prior screening.
6. Treatment at therapeutic doses/durations with any of the following within 3 months prior to randomization

   a. Natalizumab (Tysabri®) b. Cyclosporine c. Methotrexate d. Mitoxantrone e. Cyclophosphamide* f. Azathioprine g. Mycophenolate mofetil

   *Cyclophosphamide is only permitted as rescue therapy to be administered as outlined in Section 5.4.1 no earlier than the week 6 visit.
7. Severe drug allergic history or anaphylaxis to two or more food products or medicines (including known sensitivity to acetaminophen/paracetamol, diphenhydramine (cetirizine in EU) or equivalent antihistamine, and methylprednisolone or equivalent glucocorticoid).
8. Known history of a primary immunodeficiency (congenital or acquired) or an underlying condition such as human immunodeficiency virus (HIV) infection or splenectomy that predisposes the participant to infection.
9. Active malignancy or history of malignancy that was active within the last 10 years, apart from ovarian or extra-ovarian teratoma (also known as a dermoid cyst) or germ cell tumor, or squamous cell carcinoma of the skin or basal cell carcinoma of the skin, that in the opinion of the Medical Safety Monitor (MSM) would preclude enrollment due to safety concerns. Squamous cell and basal cell carcinomas should be treated with documented success of curative therapy > 3 months prior to randomization.
10. At screening (repeat testing may be conducted to confirm results within the same screening period, prior to randomization), any of the following:

    a. Total white blood count <2,500 cells/mm3 (or < 2.5 × 109/L) b. Total immunoglobulin < 600 mg/dL (or 6 µmol/L; 400 mg/dL for participants <18 years)* c. Absolute neutrophil count < 1200 cells/μL (or < 1.2 × 109/L) d. CD4 T lymphocyte count < 300 cells/µL (or < 0.3 × 109/L)

    *Baseline levels of IgG prior to first line treatments (methylprednisolone, plasmapheresis/plasma exchange) should be used to determine eligibility.
11. Active hepatitis B or C established with positive hepatitis B serology (hepatitis B surface antigen and core antigen) and/or positive hepatitis C PCR testing and confirmed by the MSM
12. Any live or attenuated vaccine within 4 weeks prior to Day 1 (administration of killed vaccines is acceptable).
13. Bacillus of Calmette and Guérin (BCG) vaccine within 1 year of enrollment.
14. History of alcohol or drug abuse that, in the opinion of the Investigator, might affect participant safety or compliance with visits or interfere with safety or other study assessments.
15. Recurrence of previously treated NMDAR encephalitis within the last 5 years, or suspicion of symptomatic untreated NMDAR encephalitis of greater than 3 months duration at the time of screening.
16. Evidence of active tuberculosis* (TB) or being at high risk for TB based on:

    a. History of active TB or untreated/incompletely treated latent TB. Participants with a history of active or latent TB who have documentation of completion of treatment according to local guidelines may be enrolled.

    b. History of recent (≤ 12 weeks of screening) close contact with someone with active TB (close contact is defined as ≥ 4 hours/week OR living in the same household OR in a house where a person with active TB is a frequent visitor).

    c. Signs or symptoms that could represent active TB by medical history or physical examination.

    d. Positive, indeterminate, or invalid interferon-gamma release assay test result at screening, unless previously treated for TB. Participants with an indeterminate test result can repeat the test once, but if the repeat test is also indeterminate, the participant is excluded.

    e. Chest radiograph, chest computed tomography or MRI scan that suggests a possible diagnosis of TB or suggests that a work-up for TB should be considered; all participants must have had lung imaging with an acceptable reading within 6 months prior to consent, or during screening.
17. Active, clinically significant (CS) infection at the time of randomization (IP administration may be delayed until recovery, if within 14-day screening window, otherwise participant may be rescreened).

Exclusion criteria are applied at time of screening and are applicable throughout the study.

* Participants will undergo QuantiFERON®-TB Gold testing or equivalent TB testing during screening as standard of care. A positive result will not exclude patients from participation; thus, enrollment should not be delayed awaiting this result. If positive, an appropriate course of anti-TB treatment will need to be documented. If results are in indeterminate, participants may still be eligible for randomization if history is not suggestive of active / latent TB and a chest x-ray shows no evidence of active or latent TB.

1.1 Additional Eligibility Considerations

The following criteria are not necessarily exclusionary but require review from the MSM to determine if a participant should be excluded due to safety concerns:

1. At screening (out of range lab values may be reviewed with the MSM to determine whether a potential participant should be excluded for safety reasons; repeat testing may be conducted to confirm results within the same screening period, prior to randomization), any of the following:

   1. Aspartate transaminase (AST) > 2.5 × age-based upper limit of normal (ULN)
   2. Alanine transaminase (ALT) > 2.5 × age-based ULN
   3. Total bilirubin > 1.5 × age-based ULN (unless due to Gilbert's syndrome)
   4. Platelet count < 75,000/μL (or < 75 × 109/L)
   5. Hemoglobin < 8 g/dL (or < 80 g/L or 5 mmol/L)
2. History of untreated hepatitis C infection. Participants who are considered cured following antiviral therapy with an HCV load below the limit of detection may be enrolled pending confirmation from the MSM that there are no safety concerns for inclusion.
3. Patients with coexistent autoantibodies should not immediately be excluded but should be reviewed with the MSM to determine eligibility.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of modified Rankin score at 16 weeks | 16 weeks
  Change in modified Rankin score (mRS) (0 to 6; 0=normal and 6=death) at 16 weeks determined by rank analyses, integrating need for rescue therapy and time to achievement of the mRS.
Inebilizumab safety measures by the number of treatment-emergent adverse events and serious adverse events | 96 weeks
  Inebilizumab safety, as measured by the number of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs)

SECONDARY OUTCOMES:
Time to mRS ≤ 2, corrected for baseline value. | 96 weeks
  Time to mRS ≤ 2, corrected for baseline value.
Clinical Assessment Scale in Autoimmune Encephalitis (CASE) Score (continuous logistic regression), corrected from baseline value to week 24 (weeks 6 and 16). | 16 weeks
  Clinical Assessment Scale in Autoimmune Encephalitis (CASE) Score (ranges of 0 to 27 with 0 being normal and 27 being worse)(continuous logistic regression), corrected from baseline value to week 24 (weeks 6 and 16).
mRS at week 6 as measured by proportional odds logistic regression/shift analysis. | 6 weeks
  mRS at week 6 as measured by proportional odds logistic regression/shift analysis.
Proportion of participants who meet the protocol-defined criteria for needing rescue therapy at week 6. | 6 weeks
  Proportion of participants who meet the protocol-defined criteria for needing rescue therapy at week 6.
Cognitive outcome at week 24 as measured by mean scaled score on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) + components of Delis-Kaplan Executive Function System (D-KEFS). | 24 weeks
  Cognitive outcome at week 24 as measured by mean scaled score on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) + components of Delis-Kaplan Executive Function System (D-KEFS).
Survival as measured by a Kaplan-Meier analysis. | 96 weeks
  Survival as measured by a Kaplan-Meier analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L Clardy, MD, PhD, Principal Investigator — University of Utah
Locations (39):
- United States (35):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph Hospital and Medical Center Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Children's Hospital of Orange County, Orange, California
  - UC Irvine, Orange, California
  - UC Davis, Sacramento, California
  - Children's Hospital Colorado Main Campus, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Ann and Robert H. Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - SUNY Downstate, Brooklyn, New York
  - Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Buffalo, Williamsville, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
- Netherlands (2):
  - Erasmus Medical University Center, Rotterdam
  - Erasmus University Rotterdam, Rotterdam
- Spain (2):
  - Hospital Clínic Barcelona, Barcelona
  - Institut d'Investigacions Biomèdiques August Pi i Sunyer (IDIBAPS), University of Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No
Data from this study will only be shared with the researchers and organizations listed in the application and consent form. Participants can opt to have their excess biosamples banked as part of an optional substudy. Any samples shared in the future will be deidentified.

REFERENCES:
- [Result] Titulaer MJ, McCracken L, Gabilondo I, Armangue T, Glaser C, Iizuka T, Honig LS, Benseler SM, Kawachi I, Martinez-Hernandez E, Aguilar E, Gresa-Arribas N, Ryan-Florance N, Torrents A, Saiz A, Rosenfeld MR, Balice-Gordon R, Graus F, Dalmau J. Treatment and prognostic factors for long-term outcome in patients with anti-NMDA receptor encephalitis: an observational cohort study. Lancet Neurol. 2013 Feb;12(2):157-65. doi: 10.1016/S1474-4422(12)70310-1. Epub 2013 Jan 3. PMID 23290630
- [Result] Gabilondo I, Saiz A, Galan L, Gonzalez V, Jadraque R, Sabater L, Sans A, Sempere A, Vela A, Villalobos F, Vinals M, Villoslada P, Graus F. Analysis of relapses in anti-NMDAR encephalitis. Neurology. 2011 Sep 6;77(10):996-9. doi: 10.1212/WNL.0b013e31822cfc6b. Epub 2011 Aug 24. PMID 21865579
- [Result] Dalmau J, Tuzun E, Wu HY, Masjuan J, Rossi JE, Voloschin A, Baehring JM, Shimazaki H, Koide R, King D, Mason W, Sansing LH, Dichter MA, Rosenfeld MR, Lynch DR. Paraneoplastic anti-N-methyl-D-aspartate receptor encephalitis associated with ovarian teratoma. Ann Neurol. 2007 Jan;61(1):25-36. doi: 10.1002/ana.21050. PMID 17262855
- [Result] Dubey D, Pittock SJ, Kelly CR, McKeon A, Lopez-Chiriboga AS, Lennon VA, Gadoth A, Smith CY, Bryant SC, Klein CJ, Aksamit AJ, Toledano M, Boeve BF, Tillema JM, Flanagan EP. Autoimmune encephalitis epidemiology and a comparison to infectious encephalitis. Ann Neurol. 2018 Jan;83(1):166-177. doi: 10.1002/ana.25131. PMID 29293273
- [Result] Dalmau J, Gleichman AJ, Hughes EG, Rossi JE, Peng X, Lai M, Dessain SK, Rosenfeld MR, Balice-Gordon R, Lynch DR. Anti-NMDA-receptor encephalitis: case series and analysis of the effects of antibodies. Lancet Neurol. 2008 Dec;7(12):1091-8. doi: 10.1016/S1474-4422(08)70224-2. Epub 2008 Oct 11. PMID 18851928
- [Result] Gresa-Arribas N, Titulaer MJ, Torrents A, Aguilar E, McCracken L, Leypoldt F, Gleichman AJ, Balice-Gordon R, Rosenfeld MR, Lynch D, Graus F, Dalmau J. Antibody titres at diagnosis and during follow-up of anti-NMDA receptor encephalitis: a retrospective study. Lancet Neurol. 2014 Feb;13(2):167-77. doi: 10.1016/S1474-4422(13)70282-5. Epub 2013 Dec 18. PMID 24360484
- [Result] Guasp M, Modena Y, Armangue T, Dalmau J, Graus F. Clinical features of seronegative, but CSF antibody-positive, anti-NMDA receptor encephalitis. Neurol Neuroimmunol Neuroinflamm. 2020 Jan 3;7(2):e659. doi: 10.1212/NXI.0000000000000659. Print 2020 Mar. PMID 31900318
- [Result] Dalmau J, Lancaster E, Martinez-Hernandez E, Rosenfeld MR, Balice-Gordon R. Clinical experience and laboratory investigations in patients with anti-NMDAR encephalitis. Lancet Neurol. 2011 Jan;10(1):63-74. doi: 10.1016/S1474-4422(10)70253-2. PMID 21163445
- [Result] Cree BAC, Bennett JL, Kim HJ, Weinshenker BG, Pittock SJ, Wingerchuk DM, Fujihara K, Paul F, Cutter GR, Marignier R, Green AJ, Aktas O, Hartung HP, Lublin FD, Drappa J, Barron G, Madani S, Ratchford JN, She D, Cimbora D, Katz E; N-MOmentum study investigators. Inebilizumab for the treatment of neuromyelitis optica spectrum disorder (N-MOmentum): a double-blind, randomised placebo-controlled phase 2/3 trial. Lancet. 2019 Oct 12;394(10206):1352-1363. doi: 10.1016/S0140-6736(19)31817-3. Epub 2019 Sep 5. PMID 31495497
- [Result] Hara M, Martinez-Hernandez E, Arino H, Armangue T, Spatola M, Petit-Pedrol M, Saiz A, Rosenfeld MR, Graus F, Dalmau J. Clinical and pathogenic significance of IgG, IgA, and IgM antibodies against the NMDA receptor. Neurology. 2018 Apr 17;90(16):e1386-e1394. doi: 10.1212/WNL.0000000000005329. Epub 2018 Mar 16. PMID 29549218
- [Result] Warikoo N, Brunwasser SJ, Benz A, Shu HJ, Paul SM, Lewis M, Doherty J, Quirk M, Piccio L, Zorumski CF, Day GS, Mennerick S. Positive Allosteric Modulation as a Potential Therapeutic Strategy in Anti-NMDA Receptor Encephalitis. J Neurosci. 2018 Mar 28;38(13):3218-3229. doi: 10.1523/JNEUROSCI.3377-17.2018. Epub 2018 Feb 23. PMID 29476014
- [Result] Hughes EG, Peng X, Gleichman AJ, Lai M, Zhou L, Tsou R, Parsons TD, Lynch DR, Dalmau J, Balice-Gordon RJ. Cellular and synaptic mechanisms of anti-NMDA receptor encephalitis. J Neurosci. 2010 Apr 28;30(17):5866-75. doi: 10.1523/JNEUROSCI.0167-10.2010. PMID 20427647
- [Result] Tuzun E, Zhou L, Baehring JM, Bannykh S, Rosenfeld MR, Dalmau J. Evidence for antibody-mediated pathogenesis in anti-NMDAR encephalitis associated with ovarian teratoma. Acta Neuropathol. 2009 Dec;118(6):737-43. doi: 10.1007/s00401-009-0582-4. PMID 19680671
- [Result] Matute C, Palma A, Serrano-Regal MP, Maudes E, Barman S, Sanchez-Gomez MV, Domercq M, Goebels N, Dalmau J. N-Methyl-D-Aspartate Receptor Antibodies in Autoimmune Encephalopathy Alter Oligodendrocyte Function. Ann Neurol. 2020 May;87(5):670-676. doi: 10.1002/ana.25699. Epub 2020 Feb 24. PMID 32052483
- [Result] Planaguma J, Leypoldt F, Mannara F, Gutierrez-Cuesta J, Martin-Garcia E, Aguilar E, Titulaer MJ, Petit-Pedrol M, Jain A, Balice-Gordon R, Lakadamyali M, Graus F, Maldonado R, Dalmau J. Human N-methyl D-aspartate receptor antibodies alter memory and behaviour in mice. Brain. 2015 Jan;138(Pt 1):94-109. doi: 10.1093/brain/awu310. Epub 2014 Nov 11. PMID 25392198
- [Result] Planaguma J, Haselmann H, Mannara F, Petit-Pedrol M, Grunewald B, Aguilar E, Ropke L, Martin-Garcia E, Titulaer MJ, Jercog P, Graus F, Maldonado R, Geis C, Dalmau J. Ephrin-B2 prevents N-methyl-D-aspartate receptor antibody effects on memory and neuroplasticity. Ann Neurol. 2016 Sep;80(3):388-400. doi: 10.1002/ana.24721. Epub 2016 Aug 2. PMID 27399303
- [Result] Malviya M, Barman S, Golombeck KS, Planaguma J, Mannara F, Strutz-Seebohm N, Wrzos C, Demir F, Baksmeier C, Steckel J, Falk KK, Gross CC, Kovac S, Bonte K, Johnen A, Wandinger KP, Martin-Garcia E, Becker AJ, Elger CE, Klocker N, Wiendl H, Meuth SG, Hartung HP, Seebohm G, Leypoldt F, Maldonado R, Stadelmann C, Dalmau J, Melzer N, Goebels N. NMDAR encephalitis: passive transfer from man to mouse by a recombinant antibody. Ann Clin Transl Neurol. 2017 Oct 3;4(11):768-783. doi: 10.1002/acn3.444. eCollection 2017 Nov. PMID 29159189
- [Result] Jones BE, Tovar KR, Goehring A, Jalali-Yazdi F, Okada NJ, Gouaux E, Westbrook GL. Autoimmune receptor encephalitis in mice induced by active immunization with conformationally stabilized holoreceptors. Sci Transl Med. 2019 Jul 10;11(500):eaaw0044. doi: 10.1126/scitranslmed.aaw0044. PMID 31292262
- [Result] Rubenstein JL, Combs D, Rosenberg J, Levy A, McDermott M, Damon L, Ignoffo R, Aldape K, Shen A, Lee D, Grillo-Lopez A, Shuman MA. Rituximab therapy for CNS lymphomas: targeting the leptomeningeal compartment. Blood. 2003 Jan 15;101(2):466-8. doi: 10.1182/blood-2002-06-1636. Epub 2002 Sep 5. PMID 12393404
- [Result] Muldoon LL, Soussain C, Jahnke K, Johanson C, Siegal T, Smith QR, Hall WA, Hynynen K, Senter PD, Peereboom DM, Neuwelt EA. Chemotherapy delivery issues in central nervous system malignancy: a reality check. J Clin Oncol. 2007 Jun 1;25(16):2295-305. doi: 10.1200/JCO.2006.09.9861. PMID 17538176
- [Result] Mei HE, Frolich D, Giesecke C, Loddenkemper C, Reiter K, Schmidt S, Feist E, Daridon C, Tony HP, Radbruch A, Dorner T. Steady-state generation of mucosal IgA+ plasmablasts is not abrogated by B-cell depletion therapy with rituximab. Blood. 2010 Dec 9;116(24):5181-90. doi: 10.1182/blood-2010-01-266536. Epub 2010 Sep 9. PMID 20829370
- [Result] Dale RC, Pillai S, Brilot F. Cerebrospinal fluid CD19(+) B-cell expansion in N-methyl-D-aspartate receptor encephalitis. Dev Med Child Neurol. 2013 Feb;55(2):191-193. doi: 10.1111/dmcn.12036. Epub 2012 Nov 14. PMID 23151040
- [Result] Makuch M, Wilson R, Al-Diwani A, Varley J, Kienzler AK, Taylor J, Berretta A, Fowler D, Lennox B, Leite MI, Waters P, Irani SR. N-methyl-D-aspartate receptor antibody production from germinal center reactions: Therapeutic implications. Ann Neurol. 2018 Mar;83(3):553-561. doi: 10.1002/ana.25173. PMID 29406578
- [Result] Chen D, Gallagher S, Monson NL, Herbst R, Wang Y. Inebilizumab, a B Cell-Depleting Anti-CD19 Antibody for the Treatment of Autoimmune Neurological Diseases: Insights from Preclinical Studies. J Clin Med. 2016 Nov 24;5(12):107. doi: 10.3390/jcm5120107. PMID 27886126
- [Result] Sanz I. Rationale for B cell targeting in SLE. Semin Immunopathol. 2014 May;36(3):365-75. doi: 10.1007/s00281-014-0430-z. Epub 2014 Apr 25. PMID 24763533
- [Result] Halliley JL, Tipton CM, Liesveld J, Rosenberg AF, Darce J, Gregoretti IV, Popova L, Kaminiski D, Fucile CF, Albizua I, Kyu S, Chiang KY, Bradley KT, Burack R, Slifka M, Hammarlund E, Wu H, Zhao L, Walsh EE, Falsey AR, Randall TD, Cheung WC, Sanz I, Lee FE. Long-Lived Plasma Cells Are Contained within the CD19(-)CD38(hi)CD138(+) Subset in Human Bone Marrow. Immunity. 2015 Jul 21;43(1):132-45. doi: 10.1016/j.immuni.2015.06.016. Epub 2015 Jul 14. PMID 26187412
- [Result] Mei HE, Wirries I, Frolich D, Brisslert M, Giesecke C, Grun JR, Alexander T, Schmidt S, Luda K, Kuhl AA, Engelmann R, Durr M, Scheel T, Bokarewa M, Perka C, Radbruch A, Dorner T. A unique population of IgG-expressing plasma cells lacking CD19 is enriched in human bone marrow. Blood. 2015 Mar 12;125(11):1739-48. doi: 10.1182/blood-2014-02-555169. Epub 2015 Jan 8. PMID 25573986
- [Result] Schuh E, Berer K, Mulazzani M, Feil K, Meinl I, Lahm H, Krane M, Lange R, Pfannes K, Subklewe M, Gurkov R, Bradl M, Hohlfeld R, Kumpfel T, Meinl E, Krumbholz M. Features of Human CD3+CD20+ T Cells. J Immunol. 2016 Aug 15;197(4):1111-7. doi: 10.4049/jimmunol.1600089. Epub 2016 Jul 13. PMID 27412413
- [Result] Herbst R, Wang Y, Gallagher S, Mittereder N, Kuta E, Damschroder M, Woods R, Rowe DC, Cheng L, Cook K, Evans K, Sims GP, Pfarr DS, Bowen MA, Dall'Acqua W, Shlomchik M, Tedder TF, Kiener P, Jallal B, Wu H, Coyle AJ. B-cell depletion in vitro and in vivo with an afucosylated anti-CD19 antibody. J Pharmacol Exp Ther. 2010 Oct;335(1):213-22. doi: 10.1124/jpet.110.168062. Epub 2010 Jul 6. PMID 20605905
- [Result] Agius MA, Klodowska-Duda G, Maciejowski M, Potemkowski A, Li J, Patra K, Wesley J, Madani S, Barron G, Katz E, Flor A. Safety and tolerability of inebilizumab (MEDI-551), an anti-CD19 monoclonal antibody, in patients with relapsing forms of multiple sclerosis: Results from a phase 1 randomised, placebo-controlled, escalating intravenous and subcutaneous dose study. Mult Scler. 2019 Feb;25(2):235-245. doi: 10.1177/1352458517740641. Epub 2017 Nov 16. PMID 29143550
- [Result] Schiopu E, Chatterjee S, Hsu V, Flor A, Cimbora D, Patra K, Yao W, Li J, Streicher K, McKeever K, White B, Katz E, Drappa J, Sweeny S, Herbst R. Safety and tolerability of an anti-CD19 monoclonal antibody, MEDI-551, in subjects with systemic sclerosis: a phase I, randomized, placebo-controlled, escalating single-dose study. Arthritis Res Ther. 2016 Jun 7;18(1):131. doi: 10.1186/s13075-016-1021-2. PMID 27267753
- [Result] Streicher K, Sridhar S, Kuziora M, Morehouse CA, Higgs BW, Sebastian Y, Groves CJ, Pilataxi F, Brohawn PZ, Herbst R, Ranade K. Baseline Plasma Cell Gene Signature Predicts Improvement in Systemic Sclerosis Skin Scores Following Treatment With Inebilizumab (MEDI-551) and Correlates With Disease Activity in Systemic Lupus Erythematosus and Chronic Obstructive Pulmonary Disease. Arthritis Rheumatol. 2018 Dec;70(12):2087-2095. doi: 10.1002/art.40656. Epub 2018 Oct 22. PMID 29956883
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Result] Balu R, McCracken L, Lancaster E, Graus F, Dalmau J, Titulaer MJ. A score that predicts 1-year functional status in patients with anti-NMDA receptor encephalitis. Neurology. 2019 Jan 15;92(3):e244-e252. doi: 10.1212/WNL.0000000000006783. Epub 2018 Dec 21. PMID 30578370
- [Result] Lim JA, Lee ST, Moon J, Jun JS, Kim TJ, Shin YW, Abdullah S, Byun JI, Sunwoo JS, Kim KT, Yang TW, Lee WJ, Moon HJ, Kim DW, Lim BC, Cho YW, Yang TH, Kim HJ, Kim YS, Koo YS, Park B, Jung KH, Kim M, Park KI, Jung KY, Chu K, Lee SK. Development of the clinical assessment scale in autoimmune encephalitis. Ann Neurol. 2019 Mar;85(3):352-358. doi: 10.1002/ana.25421. Epub 2019 Feb 10. PMID 30675918
- [Result] Lund FE, Garvy BA, Randall TD, Harris DP. Regulatory roles for cytokine-producing B cells in infection and autoimmune disease. Curr Dir Autoimmun. 2005;8:25-54. doi: 10.1159/000082086. PMID 15564716
- [Result] Lund FE. Cytokine-producing B lymphocytes-key regulators of immunity. Curr Opin Immunol. 2008 Jun;20(3):332-8. doi: 10.1016/j.coi.2008.03.003. Epub 2008 Apr 15. PMID 18417336
- [Result] Kothur K, Wienholt L, Mohammad SS, Tantsis EM, Pillai S, Britton PN, Jones CA, Angiti RR, Barnes EH, Schlub T, Bandodkar S, Brilot F, Dale RC. Utility of CSF Cytokine/Chemokines as Markers of Active Intrathecal Inflammation: Comparison of Demyelinating, Anti-NMDAR and Enteroviral Encephalitis. PLoS One. 2016 Aug 30;11(8):e0161656. doi: 10.1371/journal.pone.0161656. eCollection 2016. PMID 27575749